CLINICAL TRIAL: NCT04810481
Title: Bispectral Index and End-Tidal Anesthetic Gas Concentration in Pediatric Patients Undergoing Sevoflurane Anesthesia (BTIGER)
Brief Title: Bispectral Index and End-Tidal Anesthetic Gas Concentration in Pediatric Patients
Acronym: BTIGER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MDT20032BTIGER
Record Dates: First submitted 2021-02-25; First posted 2021-03-23 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Investigator will be blinded to the BIS value in the Standard Practice Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Practice (No Intervention): Anesthesia will be provided at the discretion of the anesthesiologist following cardiovascular variables in accordance with usual clinical indications.
- BIS Group (Active Comparator): Anesthesia will be titrated to achieve a BIS value of 45-60 during maintenance of anesthesia. Additional intervention will be provided only if the subject is in distress.
  Interventions: Device: BIS Complete Monitoring System

INTERVENTIONS:
Device: BIS Complete Monitoring System — The BIS™ complete monitoring system is a user-configurable patient monitoring system designed to monitor the hypnotic state of the brain based on the acquisition and processing of EEG signals. The BIS™ complete system processes raw EEG signals to produce a single number, called the BIS™ index, which correlates with the patient's level of hypnosis. A sensor placed on the patient's head transmits EEG signals to the BISx™ unit. The BIS™ unit filters and digitizes the signal, analyzes it for the artifact, and processes it using digital signal processing techniques to derive processed EEG parameters to a single Bispectral Index (BIS™), and finally sends the processed data to the monitor for display. The purpose of processing the EEG waveform data is to extract characteristic features from the complex signal that the BIS™ algorithm can utilize to derive BIS Index.
  Arms: BIS Group

SUMMARY:
The purpose of this study is to investigate the relationship between BIS™ values including EEG profile and anesthetic agents in the pediatric population

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational, non-invasive, randomized controlled study to collect data to compare the performance of standard practice (SP) group with the BIS™ monitoring (BIS) group. Pediatric patients between the ages of 4 to 18 years undergoing routine sevoflurane general anesthesia with an expected surgical procedure duration of greater than 30 minutes will be recruited. If the surgery is less than 15 minutes, the data will continue to be collected, but will not be included in the data analysis and the subject will be replaced with an additional subject. General surgeries including abdominal, urological, orthopedic, or ophthalmological procedures with an American Society of Anesthesiologists physical status of I - III.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Subjects (ASA physical status I or II or III) aged: 4 years to 18 years scheduled for procedures with sedation where the process of assessment will not interfere with the procedure, progress, or patient care

Exclusion Criteria:

* Has severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes, or other medical sensors
* Known neurological disorder (e.g., epilepsy, the presence of a brain tumor, a history of brain surgery, hydrocephalic disorders, depression needing treatment with anti-depressive drugs, a history of brain trauma, hemiplegia, demyelinating disorders, cerebral palsy, congenital anomalies of the brain or spinal cord, or other known neurologic disorders)
* Severe developmental delay per assessment of investigator or report of parent/guardian
* Airway abnormalities
* Pregnancy; subjects of childbearing potential will have a urine screen for pregnancy before surgery
* If the process of assessment will interfere with the procedure or the progress of the procedure
* Taking psychoactive medications
* Taking any medications that may have an impact on the Central Nervous System (CNS)
* Planned use of any regional anesthesia; a local field block is not included in this exclusion and can be used at the discretion of the anesthesia provider

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 209 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital Colorado, Aurora, Colorado
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Rutgers University, Newark, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Pittsburgh Medical Center, Children's Hospital, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Templeton TW, Alex G, Eloy JD, Stollings L, Ing RJ, Cheon EC, Belani K, Breskin I, Sebel PS, Taicher BM; BTiger Study Group. BIS Guided Titration of Sevoflurane in Pediatric Patients Undergoing Elective Surgery: A Randomized Controlled Trial. Paediatr Anaesth. 2025 Apr;35(4):277-286. doi: 10.1111/pan.15057. Epub 2025 Jan 4. PMID 39754470

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects enrolled without randomization to group (n=39) include training subject (29), screen failure (n=4), physician decision (n=2), technical problem (n=1), and other (n=3)
Groups:
- BIS Group: Anesthesia will be titrated to achieve a BIS value of 45-60 during maintenance of anesthesia. Additional intervention will be provided only if the subject is in distress.
  BIS Complete Monitoring System: The BIS™ complete monitoring system is a user-configurable patient monitoring system designed to monitor the hypnotic state of the brain based on the acquisition and processing of EEG signals. The BIS™ complete system processes raw EEG signals to produce a single number, called the BIS™ index, which correlates with the patient's level of hypnosis. A sensor placed on the patient's head transmits EEG signals to the BIS™ unit. The BIS™ unit filters and digitizes the signal, analyzes it for the artifact, and processes it using digital signal processing techniques to derive processed EEG parameters to a single Bispectral Index (BIS™), and finally sends the processed data to the monitor for display. The purpose of processing the EEG waveform data is to extract characteristic features from the complex signal that the BIS™ algorithm can utilize to derive BIS Index.
Period: Overall Study
Arm/Group | Standard Practice | BIS Group
Started | 86 | 84
Completed | 76 | 56
Not Completed | 10 | 28
Not completed — Disqualified data sets | 10 | 28

BASELINE CHARACTERISTICS:
Groups:
- BIS Group: Anesthesia will be titrated to achieve a BIS value of 45-60 during maintenance of anesthesia. Additional intervention will be provided only if the subject is in distress.
  BIS Complete Monitoring System: The BIS™ complete monitoring system is a user-configurable patient monitoring system designed to monitor the hypnotic state of the brain based on the acquisition and processing of EEG signals. The BIS™ complete system processes raw EEG signals to produce a single number, called the BIS™ index, which correlates with the patient's level of hypnosis. A sensor placed on the patient's head transmits EEG signals to the BISx™ unit. The BISx™ unit filters and digitizes the signal, analyzes it for the artifact, and processes it using digital signal processing techniques to derive processed EEG parameters to a single Bispectral Index (BIS™), and finally sends the processed data to the monitor for display. The purpose of processing the EEG waveform data is to extract characteristic features from the complex signal that the BIS™ algorithm can utilize to derive BIS Index.
- Total: Total of all reporting groups
Arm/Group | Standard Practice | BIS Group | Total
Number analyzed (Participants) | 76 | 56 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.2 (3.8) | 11.0 (3.9) | 11.1 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 47 | 26 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 16 | 32
  Not Hispanic or Latino | 57 | 38 | 95
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 14 | 34
  White | 44 | 33 | 77
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 76 | 56 | 132

OUTCOME MEASURES:

1. Primary Outcome: End-tidal Sevoflurane Concentration
Description: Average end tidal (expired) sevoflurane (ETSevo) concentration during anesthesia maintenance in pediatric patients ages 4 to 18 years. The ETSevo values from each group will be reported to show that the values are different between the BIS group when compared to the Standard Practice Group.
Time Frame: duration of maintenance of anesthesia
Population: Data in table is shown for all ages (total) and broken down by age group
Measure: Mean (Standard Deviation); unit: percent sevoflurane
Arm/Group | Standard Practice | BIS Group
Number analyzed (Participants) | 76 | 56
percent sevoflurane
  All Ages | 2.1 (0.5) | 1.8 (0.4)
  Age 4-8 years: number analyzed (Participants) | 24 | 19
  Age 4-8 years | 2.5 (0.3) | 2.1 (0.3)
  Age 9-12: number analyzed (Participants) | 23 | 18
  Age 9-12 | 2.2 (0.6) | 1.7 (0.5)
  Age 13-18: number analyzed (Participants) | 29 | 19
  Age 13-18 | 1.9 (0.5) | 1.5 (0.3)

2. Secondary Outcome: Number of Participants With Each Score on the Wong Baker Faces Scale
Description: Wong Baker FACES Scale 0-5 with 0 = No Hurt and 5 = Hurt Most
Time Frame: up to 4 hours following anesthesia administration
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Practice | BIS Group
Number analyzed (Participants) | 76 | 56
Participants
  Wong Baker FACES Scale (Highest score during PACU stay) No Hurt | 19 | 5
  Wong Baker FACES Scale (Highest score during PACU stay) Hurt Little Bit | 14 | 18
  Wong Baker FACES Scale (Highest score during PACU stay) Hurt Little More | 19 | 17
  Wong Baker FACES Scale (Highest score during PACU stay) Hurt even more | 11 | 4
  Wong Baker FACES Scale (Highest score during PACU stay) Hurt whole lot | 4 | 8
  Wong Baker FACES Scale (Highest score during PACU stay) Hurt worst | 4 | 3
  Not Reported | 5 | 1

3. Secondary Outcome: Modified Aldrete Score
Description: The Modified Aldrete Score assesses the readiness of the subject to be discharged from the post anesthesia care unit (PACU) with the higher the number correlating to the more ready a patient is to be discharged, the score range is 0-12.
Time Frame: up to 4 hours following anesthesia administration
Population: Lowest/worst timepoint reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Practice | BIS Group
Number analyzed (Participants) | 76 | 56
score on a scale | 7.3 (2.1) | 8.1 (2.0)

4. Secondary Outcome: Number of Participants With Reported Airway Reflexes
Description: Airway reflexes (e.g., coughing, choking, laryngospasm) that are common in anesthesia and not considered adverse events
Time Frame: up to 4 hours following anesthesia administration
Measure: Number; unit: participants
Arm/Group | Standard Practice | BIS Group
Number analyzed (Participants) | 76 | 56
participants
  Coughing | 13 | 4
  Choking | 0 | 0
  Laryngospasm | 0 | 0

5. Secondary Outcome: Clinical Anesthesia Assessment
Description: recorded as the number of events including movement during procedure, eye opening, hypotension, hypertension, tachycardia, bradycardia, and low oxygen saturation (SpO2) that are common in anesthesia and not considered adverse events
Time Frame: up to 4 hours following anesthesia administration
Measure: Number; unit: participants
Arm/Group | Standard Practice | BIS Group
Number analyzed (Participants) | 76 | 56
participants
  Movement during procedure | 5 | 5
  Eye opening during procedure | 3 | 3
  Hypotension during procedure | 1 | 0
  Hypertension during procedure | 1 | 0
  Tachycardia in recovery | 31 | 33
  Bradycardia in recovery | 18 | 4
  Hypotention in recovery | 39 | 19
  Hypertension in recovery | 24 | 18
  Low SPO2 in recovery | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through study exit, up to 24 hours
Arm/Group | Standard Practice | BIS Group
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/56
Serious Adverse Events (participants affected / at risk) | 1/76 | 0/56
Other Adverse Events (participants affected / at risk) | 4/76 | 3/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Practice (N=76) | BIS Group (N=56)
Pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Practice (N=76) | BIS Group (N=56)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Device Issue (Product Issues) | 0 (0) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal Abcess (Infections and infestations) | 1 (1) | 0 (0)
Endotracheal intubation complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04810481/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04810481/SAP_001.pdf